CLINICAL TRIAL: NCT00867633
Title: Observational Study of Aristolochic Acid-DNA Adduct in Urothelial Carcinoma in Taiwan
Brief Title: Aristolochic Acid-DNA Adduct in Urothelial Carcinoma in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, National Taiwan University Hospital, National Taiwan University Hospital
Other Study IDs: 200804011R
Record Dates: First submitted 2009-03-22; First posted 2009-03-24 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Urothelial Carcinoma
Keywords: urothelial carinoma; aristolochic acid; DNA; adduct
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA extracted from the resected tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Urothelial carcinoma: The DNA samples extracted from the urothelial carcinoma tissue
- RCC: the DNA sample extracted from RCC
- Non-cancer: The DNA sample extracted from the non-cancerous kidney tissue

SUMMARY:
To study the association between aristolochic acid and urothelial carcinoma in Taiwan

ELIGIBILITY:
Inclusion Criteria:

* the resected kidney tissue in the tissue bank

Exclusion Criteria:

* the patients who had been ever exposed to arsenics, rubber, chemicals, irradiation for pelvis, or received chemotherapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who received nephrectomies
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-03; Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
the incidence of aristolochic-acid DNA adduct in the samples | one week

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan